CLINICAL TRIAL: NCT04151251
Title: Mentoring Patient-Oriented Research: Sleep & Health During & After Hospital Stay
Brief Title: Inpatient Sleep Loss: Educating and Empowering Patients
Acronym: ISLEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IRB19-0169
Record Dates: First submitted 2019-10-28; First posted 2019-11-05 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Sleep

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Trained research assistants will introduce the interventions to patients, leaving the outcomes assessor and investigator only able to see results. The care provider is not part of the study decision, as the study does not affect their healthcare.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Kit Alone (Active Comparator): Patients who are not randomized into the I-SLEEP intervention will receive a sleep kit that includes an eye mask, earplugs, and headphones.They will still receive the usual standard of care provided by clinicians which includes measures to reduce unnecessary nighttime disruptions and limiting excessive noise within the hospital setting.
  Interventions: Other: Sleep Kit
- Sleep Kit + Empowerment (Experimental): A short video will be shown on iPads and a brochure will be given that both describe the importance of good sleep and how to facilitate it with good sleep hygiene.
  The video will show a few reasons why someone might not get optimal sleep while in a hospital, and offer advice to address this from a doctor. The brochure will be kept to no higher than a 6th grade reading level, considered optimal for health education materials. Text will be kept brief and to the point. To account for vision problems, we will use >12-point font & leave a large portion of each page empty. Visual Aids & graphics will be employed when possible.
  All of this is given in addition to the usual standard of care provided by clinicians.
  Interventions: Behavioral: Patient Empowerment; Other: Sleep Kit

INTERVENTIONS:
Behavioral: Patient Empowerment — Group to receive a 5 minute video about typical hospital sleep disruptions and what they can do to prevent them, as well as a brochure outlining the importance of sleep
  Arms: Sleep Kit + Empowerment
Other: Sleep Kit — Patients receive a small pouch that includes an eye mask, ear plugs, and headphones, all to be used to aid in falling/staying asleep

SUMMARY:
While many interventions have targeted hospital staff to improve sleep, few have been successful, and often suffer from limited adherence to staff protocols. Given preliminary data that suggests that empowered patients are more likely to obtain better sleep and have objectively lower noise levels in their rooms, it is plausible that partnering directly with patients can mitigate sleep loss and improve health outcomes. Patients will be randomized to receive the I-SLEEP education and empowerment program and test the effectiveness of this program on patient sleep and health outcome in the hospital and post-discharge. The aim of the project is to reduce environmental, healthcare-related, and patient-related factors that disrupt sleep of hospitalized patients by use of patient education and empowerment intervention.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the general/hospitalist medicine departments
* Stayed at least one night in hospital since admission

Exclusion Criteria:

* Admitted >72 hours ago
* Patient has been diagnosed with a sleep disorder such as narcolepsy, insomnia, or sleep apnea
* Patient was transferred from ICU or outside hospital
* Patient under strict, droplet, or airborne isolation precautions
* Unable to ambulate
* Too confused or incoherent to provide consent
* Patient cannot speak English
* Pregnancy
* Residence in a nursing home or assisted living facility
* Patient was admitted in a hospital within two weeks of current admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Karolinska Sleep Log - Sleep Times | Through stay in the hospital until discharge, usually 2-3 days
  A self-reported measure of time spent sleeping, time it took to fall asleep, etc.

SECONDARY OUTCOMES:
Frequency of Sleep Disruptions in the Hospital Setting | Through stay in the hospital until discharge, usually 2-3 days
  Administered to obtain a subjective view of typical disruptions to sleep such as bed comfort, room temperature, and pain. Items will also assess the disruptions that are caused by healthcare, such as vital signs, medication administration, and lab-work. This survey includes an item on how disruptive noise was to the patient's sleep, broken down into as many sources of hospital noise as possible.
Patients Who Report Talking to Clinicians About Their Healthcare | Through stay in the hospital until discharge, usually 2-3 days
  Measure of number of patients who advocate for their sleep by making lifestyle changes, including speaking to their clinicians to reduce nighttime disruptions
Number of nighttime disruptions to sleep | Through stay in the hospital until discharge, usually 2-3 days
  Measure of disruptions patients receive between 11 PM and 7 AM, determined by hospital hand sanitizer stations outside doors and electronic health record audits
Karolinska Sleep Log - Outcomes of Sleep | Through stay in the hospital until discharge, usually 2-3 days
  Subjective quality of sleep as determined by scales such as "On a scale of 1 to 5, with 5 being the most, how refreshed did you feel upon waking up this morning?"
Actigraphy - Objective Measure of Sleep Duration | During stay at the hospital, for a week after, and for a week three months after discharge
  Actiwatch Spectrum Pros used to determine sleep duration
Actigraphy - Objective Measure of Sleep Quality | During stay at the hospital, for a week after, and for a week three months after discharge
  Actiwatch Spectrum Pros used to determine sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Vineet Arora, MD, MAPP, Principal Investigator — Medical Researcher
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified data will be available to researchers by request

REFERENCES:
- [Background] Arora VM, Machado N, Anderson SL, Desai N, Marsack W, Blossomgame S, Tuvilleja A, Ramos J, Francisco MA, LaFond C, Leung EK, Valencia A, Martin SK, Meltzer DO, Farnan JM, Balachandran J, Knutson KL, Mokhlesi B. Effectiveness of SIESTA on Objective and Subjective Metrics of Nighttime Hospital Sleep Disruptors. J Hosp Med. 2019 Jan;14(1):38-41. doi: 10.12788/jhm.3091. PMID 30667409
- [Background] Adachi M, Staisiunas PG, Knutson KL, Beveridge C, Meltzer DO, Arora VM. Perceived control and sleep in hospitalized older adults: a sound hypothesis? J Hosp Med. 2013 Apr;8(4):184-90. doi: 10.1002/jhm.2027. Epub 2013 Mar 18. PMID 23504939
- [Derived] Mason NR, Orlov NM, Anderson S, Byron M, Mozer C, Arora VM. Piloting I-SLEEP: a patient-centered education and empowerment intervention to improve patients' in-hospital sleep. Pilot Feasibility Stud. 2021 Aug 19;7(1):161. doi: 10.1186/s40814-021-00895-z. PMID 34412696

DOCUMENTS (1):
  • Informed Consent Form (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/51/NCT04151251/ICF_000.pdf